CLINICAL TRIAL: NCT00432718
Title: Saline Instillation Before Tracheal Suctioning and the Incidence of Ventilator Associated Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Cancer, Sao Paulo (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 342/01
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2007-02-08 (Estimated); Status verified 2007-02

CONDITIONS: Mechanical Ventilation; Critically Ill Patients
Keywords: Pneumonia; Ventilator Associated Pneumonia; Prevention
MeSH Terms: conditions — Pneumonia; Pneumonia, Ventilator-Associated

INTERVENTIONS:
Procedure: Saline Instillation before Tracheal Suctioning

SUMMARY:
Compare the incidence of ventilator associated pneumonia with or without tracheal isotonic saline instillation before tracheal suctioning

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients foreseen to receive mechanical ventilation for more than 72 hours

Exclusion Criteria:

* Previous mechanical ventilation in the last month
* Mechanical ventilation for more than 6 hours before arrival at ICU,
* Contraindication to bronchoscopy and
* Be expected to die or undergo withdrawal treatment within 48 hours-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260
Dates: Start 2001-08

PRIMARY OUTCOMES:
incidence of ventilator associated pneumonia

SECONDARY OUTCOMES:
atelectasis
tube occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Caruso, MD, Principal Investigator — Intensive Care Unit - Hospital do Câncer and University of Sao Paulo Medical School
Locations (1):
- ICU Hospital do Câncer, São Paulo, São Paulo, Brazil